CLINICAL TRIAL: NCT01058213
Title: Nurse Managed Sequential Resistance Then Aerobic Training in COPD
Brief Title: Nurse Managed Sequential Strength Training and Bicycle Training in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Margaret K. Covey, Research Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NR010249
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Pulmonary rehabilitation; Resistance Training; Aerobic Training; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aerobic training alone (Active Comparator): 8 weeks of gentle chair (sham) training followed by 8 weeks of interval aerobic training on a stationary bicycle
  Interventions: Behavioral: Aerobic training
- Sequential Resistance then Aerobic Training (Experimental): 8 weeks of resistance training of the lower body followed by 8 weeks of interval aerobic training on a stationary bicycle
  Interventions: Behavioral: Resistance training; Behavioral: Aerobic training
- Concurrent resistance and aerobic training (Active Comparator): 8 weeks of gentle chair (sham) exercise followed by 8 weeks of concurrent resistance training of the lower body and interval aerobic training on a stationary bicycle
  Interventions: Behavioral: Resistance training; Behavioral: Aerobic training

INTERVENTIONS:
Behavioral: Resistance training — Supervised training will be performed on a cable exercise system (Body Solid, Forest Park, IL) using six exercises that involve concentric and eccentric muscle actions: leg press, knee flexion, knee extension, calf raise, hip adduction, hip abduction. Subjects will perform the lower extremity exercises under the direct supervision of an exercise specialist three times per week. Subjects will perform 2 sets of 8-10 repetitions at 70% of their maximum strength for 2 weeks, then will perform 2 sets of 8-10 repetitions at 80% of their maximal strength for 2 weeks, and for the next 4 weeks they will perform 3 sets of 8-10 repetitions at 80% of their maximal strength. Sets will be separated by at least a 2-3 minute rest period for multiple-joint exercises and at least 1-2 minutes for single-joint exercises. A moderate velocity of muscle contraction (~1-2 seconds for concentric and eccentric contraction) will be used.
  Arms: Concurrent resistance and aerobic training; Sequential Resistance then Aerobic Training
Behavioral: Aerobic training — Cycle ergometry training will be performed in the lab on a stationary cycle ergometer, calibrated with a 4 kg weight (Monark 828E, Varberg, Sweden). Initial work rate will be 50% of peak work rate (PWR) as tolerated and will be evaluated weekly with progressive increases targeted to achieve the highest work rate tolerated for 3-5 minutes{: wks 1-2 50% PWR, wks 3-4 60% PWR, wks 5-6 70% PWR, wks 7-8 80% PWR}. An interval training protocol will be used with subjects performing four work sets of five minutes duration separated by rest intervals of unloaded cycling lasting 2-4 minutes.

SUMMARY:
This is a 16 week exercise training program for people with severe to very severe chronic obstructive pulmonary disease (COPD). The purpose of this study is to find out if performing strength training prior to initiating exercise training on a stationary bicycle is associated with greater gains in functional status than bicycle training alone or concurrent bicycle and strength training together.

DETAILED DESCRIPTION:
Volunteers are randomly assigned to one of three groups: 1). 8 weeks of resistance (strength) training followed by 8 weeks of bicycle exercise training, 2). 8 weeks of chair exercise followed by 8 weeks of resistance (strength) training and bicycle exercise training, or 3). 8 weeks of chair exercise followed by 8 weeks of bicycle exercise training. The length of the training is 16 weeks for all 3 groups. Volunteers train 3 days per week in our lab located in the Chicagoland area and are supervised by an exercise specialist.

ELIGIBILITY:
Inclusion Criteria:

* FEV1/FVC < 70 and FEV1 < 55%,
* > 45 years of age,
* experience dyspnea with exertion,
* stable clinical condition (Stable clinical condition is defined as free of respiratory tract infections for at least two months prior to enrollment, no recent change in the color, consistency, or quantity of sputum, afebrile and no recent change in medical therapy.)

Exclusion Criteria:

* evidence of restrictive lung disease or asthma,
* acute respiratory infection,
* taking oral corticosteroids on a regular basis,
* >3 exacerbations in the previous year,
* currently participating in pulmonary rehabilitation,
* the presence of a potentially debilitating disease or the presence of a condition that would make it potentially unsafe to exercise.
* We will adhere to the American College of Sports Medicine guidelines and exclude those who do not meet their guidelines for exercise testing and training.
* Pregnant women or women who plan to become pregnant during the study.

Min Age: 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2008-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
functional capacity for aerobic exercise and for common daily activities | baseline, 16 weeks
functional reserve as measured by the reduction in breathlessness and fatigue | baseline, 16 weeks

SECONDARY OUTCOMES:
functional performance and functional capacity utilization as measured by the Functional Performance Inventory and the CHAMPS Physical Activity Scale for Older Adults | baseline, 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Margaret K Covey, PhD, RN, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Covey MK, Collins EG, Reynertson SI, Dilling DF. Resistance training as a preconditioning strategy for enhancing aerobic exercise training outcomes in COPD. Respir Med. 2014 Aug;108(8):1141-52. doi: 10.1016/j.rmed.2014.06.001. Epub 2014 Jun 11. PMID 24958605